CLINICAL TRIAL: NCT01457248
Title: Effect of Endotracheal Tube With Taper-shaped Cuff on Incidence of Postoperative Pneumonia After Aortic Surgery
Brief Title: Taper-shaped Cuff Endotracheal Tube Against Respiratory Infections
Acronym: TETRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Association pour la Recherche et la Formation en Anesthésie Analgésie Réanimation (Other)
Responsible Party: Principal Investigator, Qin Lu, Head of clinical research unit, Groupe Hospitalier Pitie-Salpetriere
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMGS-2011-1; 2011-A01038-33 (Other: Afssaps)
Record Dates: First submitted 2011-10-18; First posted 2011-10-21 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Postoperative Pneumonia
Keywords: after aortic surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endotracheal tube with taper-shaped cuff (Experimental)
  Interventions: Device: Endotracheal tube TaperGuard
- Endotracheal tube with cylindrical-shaped cuff (Active Comparator)
  Interventions: Device: Endotracheal tube Hi-Contour Brandt

INTERVENTIONS:
Device: Endotracheal tube TaperGuard — Patients are intubated by endotracheal tube with taper-shaped cuff (TaperGuard, Mallinckrodt)
  Arms: endotracheal tube with taper-shaped cuff
Device: Endotracheal tube Hi-Contour Brandt — Patients are intubated by endotracheal tube with cylindrical-shaped cuff (Hi-Contour Brandt, Mallinckrodt)
  Arms: Endotracheal tube with cylindrical-shaped cuff

SUMMARY:
The incidence of postoperative pneumonia after aortic surgery reaches 60%. In experimental lung model, endotracheal tube with taper-shaped cuff has been shown to decrease microaspiration. This effect has never been demonstrated in patients. The investigators hypothesize that use of endotracheal tube with taper-shaped cuff decreases the incidence of postoperative pneumonia in patients after aortic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Elective aortic surgery
* Admission in ICU after aortic surgery

Exclusion Criteria:

* Tracheostomized patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of first episode of postoperative pneumonia after aortic surgery | Within the first 28 days after surgery

SECONDARY OUTCOMES:
Microaspiration | Day 1 and day 2
Length of ICU stay | Participants will be followed for the duration of ICU stay, an expected average of 3 weeks
Mortality | Day 28 and day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Réanimation polyvalente, Département d'Anesthésie-Réanimation, Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Lucangelo U, Zin WA, Antonaglia V, Petrucci L, Viviani M, Buscema G, Borelli M, Berlot G. Effect of positive expiratory pressure and type of tracheal cuff on the incidence of aspiration in mechanically ventilated patients in an intensive care unit. Crit Care Med. 2008 Feb;36(2):409-13. doi: 10.1097/01.CCM.0000297888.82492.31. PMID 18007268
- [Background] Nseir S, Zerimech F, Fournier C, Lubret R, Ramon P, Durocher A, Balduyck M. Continuous control of tracheal cuff pressure and microaspiration of gastric contents in critically ill patients. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1041-7. doi: 10.1164/rccm.201104-0630OC. PMID 21836137
- [Background] Dave MH, Frotzler A, Spielmann N, Madjdpour C, Weiss M. Effect of tracheal tube cuff shape on fluid leakage across the cuff: an in vitro study. Br J Anaesth. 2010 Oct;105(4):538-43. doi: 10.1093/bja/aeq202. Epub 2010 Aug 3. PMID 20682571
- [Background] Hortal J, Giannella M, Perez MJ, Barrio JM, Desco M, Bouza E, Munoz P. Incidence and risk factors for ventilator-associated pneumonia after major heart surgery. Intensive Care Med. 2009 Sep;35(9):1518-25. doi: 10.1007/s00134-009-1523-3. Epub 2009 Jun 26. PMID 19557389